CLINICAL TRIAL: NCT01992328
Title: IVIG Treatment for Asthmatic Patients With IgG Subclass Deficiency
Acronym: IVIG
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Hae-Sim Park, Professor, Department of medicine, Ajou University School of Medicine, Ajou University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MED-CT4-12-405
Record Dates: First submitted 2013-11-11; First posted 2013-11-25 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Asthma
Keywords: Immunoglobulin G Deficiency
MeSH Terms: conditions — Asthma; IgG Deficiency | interventions — Immunoglobulins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Immune Globulin (Experimental): Immunoglobulin G Deficiency Associated with persistent asthma subtypes
  Interventions: Drug: Immune Globulin

INTERVENTIONS:
Drug: Immune Globulin — 6 months once a month intravenous immunoglobulin (400mg/kg/4weeks)
  Other Names: Immunoglobulin G Deficiency

SUMMARY:
Immunoglobulin G deficiency subtypes in patients with asthma six months once a month intravenous immunoglobulin (400mg/kg/4weeks) infection in treatment-related effect on reducing the frequency of asthma exacerbations appreciate.

DETAILED DESCRIPTION:
Patients Registration

•It is required to ensure that the patients meet the inclusion criteria for this clinical trial, are free from any items of exclusion criteria, are explained about the participation in the clinical trial along with the informed consent forms.

Procedure

•six months once a month intravenous immunoglobulin (400mg/kg/4weeks)

ELIGIBILITY:
Inclusion Criteria:

* The patient from over 16 years to under 75 years
* Patients diagnosed with asthma over six months ago
* immunoglobulin G subtypes who were diagnosed with immune deficiency
* more than 2 years Upper and lower respiratory tract infections

  , and asthma exacerbations in this regard.
* ① calculated creatinine clearance ≧ 50ml/min

  * ALT and AST <x 3 times the upper limit of normal

    * ALP <x 3 times the upper limit of normal

      * total bilirubin <x 1.5 times the upper limit of normal

Exclusion Criteria:

* within six months of the onset of the experiment who received immunoglobulin therapy
* immune globulin for those with a history of hypersensitivity reactions
* six months ago, another clinical trial participants.
* Systemic steroids and immunomodulators, such as asthma control that may affect the resources required drug administration.
* pregnant or lactating women.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-12; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Infection rate | 6months
  6 months after treatment compared to before treatment 6 months

SECONDARY OUTCOMES:
lung funtion | 6 months
  - Lung function (FEV1) compared
steroid | 6 months af
  - Systemic steroid dose and the number of uses
antibiotic | 6months
  - The frequency and duration of antibiotic
asthma syptoms | 6months
  - The frequency of asthma exacerbations
Questionnaire | 6months
  - Asthma Quality of Life (AQOL)
Questionnair | 6months
  - Asthma control score (K-ACT)
IgG subclass | 6months
  - Before and after treatment serum IgG subclass
Cytokines | 6months
  - Cytokines serum levels before and after treatment
adverse events | 6months
  - The frequency of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: hae-sim park, Principal Investigator — Department of medicine, Ajou University School of Medicine